CLINICAL TRIAL: NCT06870812
Title: Rapid Evacuation and Access of Cerebral Hemorrhage Trial
Acronym: REACH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: The Marcus Foundation (Other)
Responsible Party: Principal Investigator, Alex Hall, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00008310; 2025P011235 (Other: Emory IRB)
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Stroke Hemorrhagic
Keywords: Intracerebral hemorrhage; minimally invasive surgery; Blood clot
MeSH Terms: conditions — Hemorrhagic Stroke; Cerebral Hemorrhage; Thrombosis | interventions — Practice Management, Medical; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical management (MIPS) plus medical management (Experimental): Participants randomized to surgical management will follow the Medical Manual of the Clinical Standardization Guidelines (CSG) before and after surgery.
  Interventions: Procedure: Surgical management; Other: Medical Management
- medical management. (Active Comparator): Participants randomized to the medical management alone will be treated according to the Clinical Standardization Guidelines (CSG).
  Interventions: Other: Medical Management

INTERVENTIONS:
Procedure: Surgical management — Following randomization into the surgical arm, a competency-trained neurosurgeon will perform the MIPS for clot evacuation with strict adherence to the Surgical Manual of the CSG. Image interpretation, patient position, anesthetic plan, stereotactic navigation registration, exoscopic positioning, access, optics, resection, and hemostasis are detailed in the Surgical Manual of the CSG.
  The OR arrival time should occur <24 hours from the last known normal (LKN) with a goal of arrival in less than 8 hours from the last known normal.
  Other Names: Early minimally invasive parafascicular surgery (MIPS)
  Arms: Surgical management (MIPS) plus medical management
Other: Medical Management — Following randomization into the medical arm patients will be treated following the Medical Manual of the CSG. The Medical Manual has been adapted by the REACH Executive Committee (REC) from the current American Heart Association (AHA) and American Stroke Association (ASA) Guidelines for the Management of Spontaneous Intracerebral Hemorrhage. Whenever clinically feasible, the CSG should be followed as it represents a template for the care of these subjects.
  The Medical Manual details specialty level of care, including intensive care placement, blood pressure control, hemostasis and coagulopathy, anemia, deep venous thrombosis and pulmonary embolism prophylaxis/treatment, glucose management, temperature management, seizure prophylaxis, intracranial pressure monitoring and management, intraventricular hemorrhage (IVH)/obstructive hydrocephalus management, cerebral edema, decompressive hemicraniectomy, nutritional support, respiratory support, and comfort care.
  Other Names: Standard of Care (SOC)

SUMMARY:
The main purpose of this study is to compare patients with a deep bleed in the brain undergoing surgery to patients receiving routine medical care. The standard treatment involves admission to the Intensive Care Unit (ICU) with close monitoring and blood pressure control. It also includes other medical (non-surgical) treatments to prevent more bleeding or another stroke. Sometimes, doctors will recommend surgery to remove the blood if medical treatment alone is not successful.

There is evidence that doing minimally invasive surgery early-using a small opening in the skull to remove blood-may help some patients. Researchers aim to understand whether this surgery is better than current medical treatment, which may include surgeries to relieve pressure on the brain in some cases. This study, called REACH, is comparing usual medical care to early minimally invasive surgery so doctors can know which is better for patients.

DETAILED DESCRIPTION:
The REACH trial, which stands for Rapid Evacuation and Access of Cerebral Hemorrhage Trial, is a medical research study aimed at finding better ways to treat people who have had a specific type of stroke called an intracerebral hemorrhage. This type of stroke happens when a blood vessel bursts and causes bleeding in the brain.

Traditionally, treating this kind of stroke has been challenging, and the best approach is not always clear. Recently, trials have shown that minimally invasive surgery to remove the clot caused by bleeding improves outcomes and decreases death when the blood is located closer to the surface of the skull. The REACH trial is testing the same minimally invasive surgery to remove the blood clot caused by the bleeding in a deeper part of the brain. The goal is to see if this approach can improve recovery and outcomes for patients compared to standard medical care.

In simple terms, the REACH trial is trying to find out if using a less invasive surgical technique can help people recover better and faster after a bleeding stroke in the deeper part of the brain.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Pre-randomization head CT demonstrating an acute, spontaneous, anterior basal ganglia primary intracerebral hemorrhage (ICH) (the anterior basal ganglia include the caudate, putamen, and pallidum to the capsula externa and excludes the thalamus)
* ICH volume between 20 - 80 mL as calculated by an approved and standardized volumetric measurement
* Study intervention can reasonably be initiated within 24 hours after the onset of stroke symptoms. If the onset is unclear, then the onset will be considered the time that the subject was last known to be well.
* Glasgow Coma Score (GCS) 5 - 14
* Historical Modified Rankin Score 0 or 1

Exclusion Criteria:

* Ruptured aneurysm, arteriovenous malformation (AVM), vascular anomaly, Moyamoya disease, venous sinus thrombosis, mass or tumor, hemorrhagic conversion of an ischemic infarct, recurrence of a recent (less than 1 year) ICH, as diagnosed with radiographic imaging
* NIH Stroke Scale (NIHSS) less than or equal to 5
* Bilateral fixed dilated pupils
* Extensor motor posturing
* Intraventricular extension of the hemorrhage is visually estimated to involve greater than 50% of either of the lateral ventricles
* Primary thalamic ICH or basal ganglia hemorrhage with involvement > 25% of thalamus
* Infratentorial intraparenchymal hemorrhage including midbrain, pontine, or cerebellar
* Use of anticoagulants that cannot be rapidly reversed (i.e., criteria is met if investigators are confident that clinically significant coagulopathy is not present after targeted correction)
* Evidence of active bleeding involving a retroperitoneal, gastrointestinal, genitourinary, or respiratory tract site
* Uncorrected coagulopathy or known clotting disorder
* Known platelet count less than 75,000 or known international normalized ratio (INR) greater than 1.4 after correction
* Patients requiring long-term anti-coagulation that needs to be initiated less than or equal to 5 days from initial ICH
* End-stage renal disease
* Patients with a mechanical heart valve
* End-stage liver disease
* History of drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Positive urine or serum pregnancy test in female subjects without documented history of surgical sterilization or post-menopausal
* Known life expectancy of less than 6 months before ICH
* No reasonable expectation of recovery, do-not-resuscitate (DNR), or comfort measures only before randomization
* Participation in a concurrent interventional medical investigation or clinical trial. Patients in non-interventional/observational studies are eligible
* Inability or unwillingness of the subject or legal guardian/representative to give written informed consent
* Homelessness or inability to meet follow-up requirements

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Score on the modified Rankin Scale (mRS) at | 180 days after randomization
  The mRS is a seven-level ordinal scale that ranges from 0 (no symptoms) to 6 (death).

SECONDARY OUTCOMES:
Hospital mortality | Up to 14 days (average hospital stay)
  Mortality rate during hospitalization will be calculated.
All-cause mortality at discharge from the initial hospitalization | 30 days after randomization
  All-cause mortality rate will be calculated.
Change in hematoma volume | Baseline and up to 36 hours post-randomization
  The change in hematoma volume from the initial to the follow-up neuroimaging for surgical management versus medical management.
Post-operative rebleeding associated with neurologic deterioration | Up to 36 hours post-randomization
  Post-operative rebleeding associated with neurologic deterioration (defined as a growth in hematoma volume between the initial CT and follow-up neuroimaging and an increase of 4 or more points on the NIH stroke scale or a decrease of up to 2 points on the GCS that was not explained by planned medical interventions [e.g., sedatives, analgesics, and procedures]).
  *This outcome applies to the surgery group only.
Serious adverse events | 180-days post-randomization
  All adverse events will be recorded f after randomization until the final follow-up visit.
Number of participants who required a decompressive hemicraniectomy | Up to 14 days (average stay in the hospital)
  Number of participants who required a decompressive hemicraniectomy in each group during initial hospitalization.
Intensive care unit (ICU) length-of-stay (LoS) | Up to 7 days (average stay in ICU)
  Total number of days spent in ICU
Duration of mechanical ventilation between groups | Up to 7 days (average ICU stay)
  Duration that patients required mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Alex Hall, DHSc, Principal Investigator — Emory University; Gustavo Pradilla, MD, Principal Investigator — Emory University; Jonathan Ratcliff, MD, Principal Investigator — Emory University
Locations (7):
- United States (7):
  - Baptist Health Jacksonville FL, Jacksonville, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital (EUH), Atlanta, Georgia
  - Rush University, Chicago, Illinois
  - Endeavor Health, Northshore, Evanston, Illinois
  - SUNY Upstate Medical University, Syracuse, New York

IPD SHARING:
Plan to Share IPD: Yes
The research team will share de-identified data upon reasonable request and approval by the Executive Committee no earlier than one year after the primary manuscript is published.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available one year after the publication of the primary manuscript.
Access Criteria: One year after the publication, academic institutions or industry researchers may submit requests to contribute to tertiary, meta, and other exploratory analyses and publications to the publications committee, provided they include a methodologically sound proposal. Proposals should be sent to REACHTRIAL@emory.edu. Data Transfer Agreements may be required.